CLINICAL TRIAL: NCT03390439
Title: Treatment of Atrofic Striae With Percutaneous Collagen Induction Therapy Versus Fractional Nonablative Laser: a Randomized Trial
Brief Title: Treatment of Atrofic Striae With Percutaneous Collagen Induction Therapy Versus Fractional Nonablative Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other); MTO Importadora e Distribuidora (Unknown); Vydence Medical (Unknown); Aché Laboratórios Farmacêuticos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 47639415.1.0000.5327
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2017-06

CONDITIONS: Striae Distensae
Keywords: Striae alba; Microneedling; Fractional nonablative laser; dermaroller; Nd-yap 1340nm laser; Percutaneous Collagen Induction Therapy
MeSH Terms: conditions — Striae Distensae | interventions — Lasers; Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Each patient will have the abdomen divided equally. Each segment of the abdomen will be randomized using the Excel 2013 program to receive laser or microneedle treatment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical evaluators will evaluate the photos after the treatments blindly for which type of treatment applied.
  Evaluators of skin biopsies will be blinded to what type of treatment is applied and for pre-treatment and post-treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nd-Yap 1340nm laser (Active Comparator): The randomly assigned segment of the abdomen will receive 5 sessions with monthly intervals of Nd-yap 1340nm laser.
  Interventions: Device: Nd-Yap 1340nm laser
- Microneedling (Experimental): The randomly assigned segment of the abdomen will receive 5 sessions with monthly intervals of dermaroller 2,5mm.
  Interventions: Device: Microneedling

INTERVENTIONS:
Device: Nd-Yap 1340nm laser — Each part of the abdomen will be treated with a therapeutic modality. The ND-yap 1340-nm laser will be used in the following parameters: 90 mtz / cm2 nozzle, 90 mJ / mtz power, 2.5 Hz frequency, 3 ms pulse duration, 1 pass.
  Other Names: Nonablative Fractional Laser
  Arms: Nd-Yap 1340nm laser
Device: Microneedling — In the other segment of the abdomen, the dermaroller 2.5 mm will be applied, with ten to fifteen passes in the same direction and at least four crosses in the rolling areas.
  Other Names: Dermaroller; Percutaneous Collagen Induction Therapy
  Arms: Microneedling

SUMMARY:
As atrophic striae are common dermatological conditions. Various therapeutic modalities have been employed in the treatment of striae distensae, mainly in striae rubra. There are few studies that include the treatment of striae alba.

The non-ablative fractionated laser and, more recently, microneedling are two distinct treatments, but they are widely used in dermatologist practice.

The present randomized clinical trial is aimed at evaluating and evaluating the response of microneedle and fractional non-ablative laser Nd-yap 1340 in the treatment of abdominal striae alba.

DETAILED DESCRIPTION:
Twenty patients will be treated at the dermatologic clinic of the Hospital de Clínicas de Porto Alegre (HCPA). Each patient will be treated with laser and microneedle at the same time, being applied a therapeutic procedure in each part of the abdomen (divided lengthwise and in equal parts). Each part of the abdomen will be randomized for the treatment of laser or microneedling with the help of the Excel 2013 program. The investigator responsible for procedures and patients are the only ones with unblinded assessment in relation to the side of each treatment. There will be 5 sessions with monthly intervals of the proposed treatments. The ND-yap 1340-nm laser will be used, and in the other segment of the abdomen, the dermaroller 2.5 mm was applied. Photographic records of patients will be performed at pre-treatment and 1 month after the third and fifth sessions. The questionnaires will be applied to assess the quality of life in dermatology DLQI (Dermatology Life Quality Index). Two independent and blind evaluators for the type of treatment will apply in the Global Aesthetic Scale (GAIS) in the evaluation of photographic records. Cutaneous biopsies for histopathological evaluation will be performed with a punch 3 mm of each part of the abdomen at pretreatment. Two experienced pathologists will evaluate the measurements of the epidermis and the collagen and elastic fibers of the skin.

ELIGIBILITY:
Inclusion Criteria:

* female patients,
* age 18 and over;
* presenting with abdominal striae rubra diagnosed after clinical examination;
* patients with weight stability in the last four months;
* patients with Fitzpatrick III or IV phototype.

Exclusion Criteria:

* pregnant women;
* childbirth for less than 12 months;
* history of keloid scars;
* presence of localized or systemic infection;
* presence of immunosuppression;
* use of photosensitizing medications;
* use of systemic steroids;
* use of oral isotretinoin in the last 12 months;
* history of diseases of collagen or elastic fibers;
* hypersensitivity to infiltrative or topical anesthetics;
* patients who have been treated for striae distensae in the last year;
* presence of sun exposure during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Clinical response in abdominal alba striae after the therapies | 6 months
  Clinical response to microneedle treatment and nonablative fractional laser treatment without abdominal alba striae (GAIS scale). The GAIS scale is a non-numerical scale divided into 5 categories of clinical response: very much improved, much improved, improved, no changed and worse.

SECONDARY OUTCOMES:
Clinical response to microneedle treatment and nonablative fractional laser treatment | 4 months
  Clinical response to microneedle treatment and nonablative fractional laser treatment without abdominal alba striae (GAIS scale). The GAIS scale is a non-numerical scale divided into 5 categories of clinical response: very much improved, much improved, improved, not changed and worse.
Histopatological response in abdominal striae alba after the therapies | 4 months
  Histopathological evaluation of the thickness of the epidermis, as collagen and elastic (picrosirius stain, orcein stain)
Histopatological response in abdominal striae alba after the therapies | 6 months
  Histopathological evaluation of the thickness of the epidermis, as collagen and elastic (picrosirius stain, orcein stain)
The tolerability and incidence of adverse effects during the therapies | 1 month
  To assess the tolerability and the incidence of immediate and late adverse effects (pain, skin erythema, pruritus) for both techniques
The tolerability and incidence of adverse effects during the therapies | 2 months
  To assess the tolerability and the incidence of immediate and late adverse effects (pain, skin erythema, pruritus) for both techniques
The tolerability and incidence of adverse effects during the therapies | 3 months
  To assess the tolerability and the incidence of immediate and late adverse effects (pain, skin erythema, pruritus) for both techniques
The tolerability and incidence of adverse effects during the therapies | 4 months
  To assess the tolerability and the incidence of immediate and late adverse effects (pain, skin erythema, pruritus) for both techniques
The tolerability and incidence of adverse effects during the therapies | 5 months
  To assess the tolerability and the incidence of immediate and late adverse effects (pain, skin erythema, pruritus) for both techniques
The impact on the quality of life provided by the striae distensae | Pre-treatment (first day of the evaluation)
  To evaluate the impact on the quality of life (DLQI) provided by the striae. It is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions.The DLQI is the most frequently used instrument in studies of randomised controlled trials in dermatology.
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  0-1: no effect at all on patient's life 2-5: small effect on patient's life 6-10: moderate effect on patient's life 11-20: very large effect on patient's life 21-30:extremely large effect on patient's life
The impact on the quality of life provided by the striae distensae | 4 months
  To evaluate the impact on the quality of life (DLQI) provided by the striae. It is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions.The DLQI is the most frequently used instrument in studies of randomised controlled trials in dermatology.
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  0-1: no effect at all on patient's life 2-5: small effect on patient's life 6-10: moderate effect on patient's life 11-20: very large effect on patient's life 21-30:extremely large effect on patient's life.
The impact on the quality of life provided by the striae distensae | 6 months
  To evaluate the impact on the quality of life (DLQI) provided by the striae. It is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions.The DLQI is the most frequently used instrument in studies of randomised controlled trials in dermatology.
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  0-1: no effect at all on patient's life 2-5: small effect on patient's life 6-10: moderate effect on patient's life 11-20: very large effect on patient's life 21-30:extremely large effect on patient's life.

CONTACTS AND LOCATIONS:
Overall Officials: Tania F Cestari, Dr, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Ana Paula Naspolini, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Himdani S, Ud-Din S, Gilmore S, Bayat A. Striae distensae: a comprehensive review and evidence-based evaluation of prophylaxis and treatment. Br J Dermatol. 2014 Mar;170(3):527-47. doi: 10.1111/bjd.12681. PMID 24125059
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Yang YJ, Lee GY. Treatment of Striae Distensae with Nonablative Fractional Laser versus Ablative CO(2) Fractional Laser: A Randomized Controlled Trial. Ann Dermatol. 2011 Nov;23(4):481-9. doi: 10.5021/ad.2011.23.4.481. Epub 2011 Nov 3. PMID 22148016
- [Background] Geronemus RG. Fractional photothermolysis: current and future applications. Lasers Surg Med. 2006 Mar;38(3):169-76. doi: 10.1002/lsm.20310. PMID 16532440
- [Background] de Angelis F, Kolesnikova L, Renato F, Liguori G. Fractional nonablative 1540-nm laser treatment of striae distensae in Fitzpatrick skin types II to IV: clinical and histological results. Aesthet Surg J. 2011 May;31(4):411-9. doi: 10.1177/1090820X11402493. PMID 21551432
- [Background] Cachafeiro T, Escobar G, Maldonado G, Cestari T, Corleta O. Comparison of Nonablative Fractional Erbium Laser 1,340 nm and Microneedling for the Treatment of Atrophic Acne Scars: A Randomized Clinical Trial. Dermatol Surg. 2016 Feb;42(2):232-41. doi: 10.1097/DSS.0000000000000597. PMID 26845539
- [Background] Park KY, Kim HK, Kim SE, Kim BJ, Kim MN. Treatment of striae distensae using needling therapy: a pilot study. Dermatol Surg. 2012 Nov;38(11):1823-8. doi: 10.1111/j.1524-4725.2012.02552.x. Epub 2012 Aug 22. PMID 22913429
- [Background] Hexsel D, Soirefmann M, Porto MD, Schilling-Souza J, Siega C, Dal'Forno T. Superficial dermabrasion versus topical tretinoin on early striae distensae: a randomized, pilot study. Dermatol Surg. 2014 May;40(5):537-44. doi: 10.1111/dsu.12460. Epub 2014 Feb 26. PMID 24612027
- [Background] Zeitter S, Sikora Z, Jahn S, Stahl F, Strauss S, Lazaridis A, Reimers K, Vogt PM, Aust MC. Microneedling: matching the results of medical needling and repetitive treatments to maximize potential for skin regeneration. Burns. 2014 Aug;40(5):966-73. doi: 10.1016/j.burns.2013.12.008. Epub 2014 Feb 7. PMID 24513133
- [Background] Aust MC, Fernandes D, Kolokythas P, Kaplan HM, Vogt PM. Percutaneous collagen induction therapy: an alternative treatment for scars, wrinkles, and skin laxity. Plast Reconstr Surg. 2008 Apr;121(4):1421-1429. doi: 10.1097/01.prs.0000304612.72899.02. PMID 18349665
- [Derived] Naspolini AP, Boza JC, da Silva VD, Cestari TF. Efficacy of Microneedling Versus Fractional Non-ablative Laser to Treat Striae Alba: A Randomized Study. Am J Clin Dermatol. 2019 Apr;20(2):277-287. doi: 10.1007/s40257-018-0415-0. PMID 30618025